CLINICAL TRIAL: NCT03103906
Title: A Randomized, Evaluator-blind, Single-center and Two Arm Clinical Study Designed to Evaluate the Local Tolerance and Cosmetic Efficacy of a Topical Skin Care Formulation in Healthy Female Subjects With Mild to Advanced Photo-damaged Facial Skin Who Have Undergone a 70% Glycolic Acid Facial Peel Procedure
Brief Title: Evaluation of the Cosmetic Benefit of a Skin Cream in Healthy Females With Mild to Advanced Photo-damaged Facial Skin Who Have Undergone a Glycolic Acid Facial Peel Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207213
Record Dates: First submitted 2017-03-24; First posted 2017-04-06 (Actual); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Skin Care
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Test Product) (Experimental): Participants will apply test product (approximately 0.6-1 grams (g)) to full face topically twice daily (morning and evening) after cleansing. All participants will be instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
  Interventions: Other: Cream (Test product); Other: Cleanser (Reference Product); Other: Sunscreen (Reference Product)
- Group 2 (No Treatment) (Other): Participants will wet face with water and work a small amount of facial cleanser (approximately 0.6-1 g) into lather. Participants will massage topically onto wet skin and rinse with water twice daily (morning and evening). After cleansing, participants will apply a pea-sized quantity (approximately 0.6-1 g) of the sunscreen in the morning and at lunchtime.
  Interventions: Other: Cleanser (Reference Product); Other: Sunscreen (Reference Product)

INTERVENTIONS:
Other: Cream (Test product) — Moisturizing cream with SPF (Sun protecting factor) 20
  Arms: Group 1 (Test Product)
Other: Cleanser (Reference Product) — Moisturizing facial cleanser
Other: Sunscreen (Reference Product) — SPF 50 sunscreen

SUMMARY:
Evaluation of the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female participants with mild to advanced photo-damaged facial skin who have undergone a 70% Glycolic Acid facial peel procedure.

DETAILED DESCRIPTION:
A randomized, evaluator-blind, single-center and two-arm clinical study designed to evaluate the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female participants with mild to advanced photo-damaged facial skin who have undergone a 70% Glycolic Acid facial peel procedure.

ELIGIBILITY:
Inclusion Criteria

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Females aged between 30 and 60 years inclusive.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination.
* Willingness to actively participate in the study and to attend all scheduled visits.
* Skin type: a) Fitzpatrick phototype II-IV. b) Participants with Glogau photoaging type II-III.
* Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone or injectable progestogen or implants of levonorgestrel or estrogenic vaginal ring or percutaneous contraceptive patches or intrauterine device or intrauterine system or double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) or male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant.

Exclusion Criteria

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* a) Active skin disease or open wound in the test area b)Medical history of using a medicated acne treatment (e.g. Benzoyl Peroxide, Clindamycin, isotretinoin) within the last 24 months, c) Medical history of dysplastic nevi or melanoma, d) Preexisting inflammatory dermatoses such as psoriasis, atopic dermatitis, e) Moles, tattoos, scars, irritated skin, hairs, etc. at the test area that could, in the opinion of the investigator, influence the investigation, e) Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines within 7 days prior to screening and/or throughout the entire course of the study, g) Systemic use of over-the-counter (OTC) analgesics or anti-inflammatory drugs 24 hours prior to screening, h) Systemic use of any photosensitizing medication 2 weeks prior to screening, i) Intense sun exposure, UV-treatments or tanning salon visit within two weeks prior to screening, j)One of the following illnesses that might require regular systemic medication: Insulin-dependent diabetes, cancer k) One of the following illnesses if not medicated: Asthma, hypertension, l) Medical history of abnormal response to sunlight, m)Participants with a history of mental illness, n) Ocular surgery within the last 12 months, o) Ocular trauma, infection or inflammation within the last 3 months, p) Active blepharitis, conjunctivitis, uveitis, q) Any ocular pathology requiring topical ocular treatment within the last 1 month, r) Ocular laser within the last 3 months, s) Aesthetic, cosmetic or dermatological treatment in the treatment area (face), including the use of skin tone lightning products, within the last 3 months, t) Use of facial scrubs, depilatory creams, waxing and/or bleaching within the last 2 weeks prior to screening, u) Microdermabrasion and/or laser hair removal within the last 4 weeks prior to screening, and v) Medical history of Herpes Simplex (Cold Sores).
* a) Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients, b) Documented allergies to cosmetic products or study ingredients.
* a) Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit, b) Previous participation in this study.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* a) Required to work outside during daylight hours over the duration of the study, b) Required or otherwise intending to spend prolonged periods of time outside during daylight hours over the duration of the study (e.g. holiday, sunbathing, and gardening).
* A score of "Severe" for any Dermatologist or Participant Self-Assessed endpoint at any time for the study material sensitivity test.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in Brazil.
Pre-assignment Details: A total of 141 participants were screened, out of which 106 participants were enrolled in the study. 35 participants were not enrolled as 30 did not met study criteria, 2 had adverse event and 3 were lost to follow up. Out of 106, 82 participants were randomized and 24 were not randomized because of other reasons (unspecified).
Groups:
- Group 1 (Test Product): Participants were instructed to apply test product (approximately 0.6-1 g[gram]) to full face topically twice daily (morning and evening) after cleansing for a total of 14 consecutive days. All participants were instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
- Group 2 (No Test Product): Participants were instructed to use the facial cleanser twice-daily during the morning and evening, and to apply the sunscreen in the morning and at lunchtime for a total of 14 consecutive days.
Period: Overall Study
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Started | 40 | 42
Completed | 36 | 39
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants with at least one application of product (i.e. test product for participants in Group 1 or sunscreen for participants in Group 2).
Groups:
- Group 1 (Test Product): Participants were instructed to apply test product (approximately 0.6-1 g) to full face topically twice daily (morning and evening) after cleansing for a total of 14 consecutive days. All participants were instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product) | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (8.41) | 46.5 (8.04) | 46.4 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 77
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Evaluator (Dermatologist) Global Assessment (EGA) Score for Well Tolerance of Product 14 Days Post-Procedure
Description: The Dermatologist assessed the local tolerance of the post-procedure skin care regimen in context of the expected effects of the procedure for each participant using the scale below: 0 - Product regimen was well tolerated (No clinically significant worsening of the expected signs/symptoms of the procedure. No new signs/symptoms manifest during product use) and 1 - Product regimen was not well tolerated (Clear, clinically relevant worsening of the severity or frequency of expected signs/symptoms of the procedure and/or any occurrence of new, unexpected signs/symptoms during product use). The Dermatologist drawn assessment on the total set of clinical and participant self-assessment data for each participant.
Time Frame: 14 days after completion of the facial peel procedure
Population: Safety population included all participants with at least one application of product (i.e. test product for participants in Group 1 or sunscreen for participants in Group 2). Number of participants analyzed are the part of safety population analyzed for this outcome 14 days post-procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 36 | 39
Participants | 36 | 38
Statistical Analysis 1: Comparison: Group 1 (Test Product) vs Group 2 (No Test Product); Test type: Other; p = 0.3334, Chi-squared; Difference in proportion = 2.56, 95% CI 2-sided [-19.99 to 25.07]

2. Secondary Outcome: Change From Baseline in Total Score of Dermatologist Assessment Score
Description: Participants scored for all domains of Dermatologist Assessment Score using scale of 0 to 3. Erythema (0=None-No evidence of erythema present, 1=Mild-Slight red coloration, 2=Moderate-Definite redness, 3=Severe-Marked erythema, bright red to dusky dark red), Dryness (0=None-No dryness, 1=Mild-Barely perceptible, fine scales or flakes present to limited areas of the test site, 2=Moderate-Fine scales or flakes generalized to all areas of the test site, 3=Severe -Scaling & peeling of skin over all areas of the test site), Desquamation (0=None-No evidence of desquamation/peeling, 1=Mild-Barely perceptible scaling; evident only on scratching, 2=Moderate-Minimal scaling, adherent to the skin, 3=Severe -Moderate scaling, loosely adherent to the skin & easily removable), Edema (0=None-No edema present, 1=Mild-Barely perceptible edema present, 2=Moderate-Definite edema present, 3=Severe Marked/pronounced edema present). Total score as 0 to 12, higher scores represent less local tolerance.
Time Frame: At baseline (60 minutes post procedure but prior to any test product application), 180 minutes, 1 day, 2 days, 3 days, 7 days and 14 days after completion of the facial peel procedure
Population: Safety population included all participants with at least one application of product (i.e. test product for participants in Group 1 or sunscreen for participants in Group 2). Number of participants analyzed are the part of safety population evaluated for this outcome at specific time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
score on a scale
  At Baseline | 0.49 (0.651) | 0.73 (0.816)
  Change from baseline at 180 min. post procedure | -0.22 (0.479) | -0.25 (0.494)
  Change from baseline at Day 1 post procedure | 0.24 (0.925) | 0.18 (0.984)
  Change from baseline at Day 2 post procedure: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 2 post procedure | 0.14 (0.723) | 0.23 (0.862)
  Change from baseline at Day 3 post procedure: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 3 post procedure | 0.11 (0.950) | 0.50 (1.155)
  Change from baseline at Day 7 post procedure: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 7 post procedure | -0.17 (0.655) | -0.33 (0.701)
  Change from baseline at Day 14 post procedure: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 14 post procedure | -0.25 (0.937) | -0.51 (0.914)

3. Secondary Outcome: Change From Baseline in Individual Dermatologist Assessment Scores of Erythema, Dryness, Desquamation and Edema
Description: Participants scored for all domains of Dermatologist Assessment Score using scale of 0 to 3. Erythema (0=None-No evidence of erythema present, 1=Mild-Slight red coloration, 2=Moderate-Definite redness, 3=Severe-Marked erythema, bright red to dusky dark red), Dryness (0=None-No dryness, 1=Mild-Barely perceptible, fine scales or flakes present to limited areas of the test site, 2=Moderate-Fine scales or flakes generalized to all areas of the test site, 3=Severe -Scaling & peeling of skin over all areas of the test site), Desquamation (0=None-No evidence of desquamation/peeling, 1=Mild-Barely perceptible scaling; evident only on scratching, 2=Moderate-Minimal scaling, adherent to the skin, 3=Severe -Moderate scaling, loosely adherent to the skin & easily removable), Edema (0=None-No edema present, 1=Mild-Barely perceptible edema present, 2=Moderate-Definite edema present, 3=Severe Marked/pronounced edema present). Higher scores represent less local tolerance.
Time Frame: At baseline (60 minutes. post procedure but prior to any test product application) and 180 minutes, 1 day, 2 days, 3 days, 7 days and 14 days after completion of the facial peel procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
score on a scale
  Erythema: At Baseline | 0.32 (0.530) | 0.48 (0.640)
  Erythema: Change from baseline at 180 minutes | -0.11 (0.393) | -0.23 (0.480)
  Erythema: Change from baseline at Day 1 | -0.03 (0.552) | -0.15 (0.700)
  Erythema: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Erythema: Change from baseline at Day 2 | -0.17 (0.378) | -0.23 (0.620)
  Erythema: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Erythema: Change from baseline at Day 3 | -0.14 (0.593) | -0.10 (0.744)
  Erythema: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Erythema: Change from baseline at Day 7 | -0.25 (0.554) | -0.41 (0.595)
  Erythema: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Erythema: Change from baseline at Day 14 | -0.19 (0.668) | -0.36 (0.707)
  Dryness: At Baseline | 0.14 (0.347) | 0.18 (0.385)
  Dryness: Change from baseline at 180 minutes | -0.08 (0.277) | 0.05 (0.316)
  Dryness: Change from baseline at Day 1 | 0.16 (0.501) | 0.20 (0.464)
  Dryness: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Dryness: Change from baseline at Day 2 | 0.14 (0.593) | 0.30 (0.516)
  Dryness: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Dryness: Change from baseline at Day 3 | 0.08 (0.554) | 0.33 (0.526)
  Dryness: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Dryness: Change from baseline at Day 7 | 0.06 (0.410) | 0.05 (0.456)
  Dryness: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Dryness: Change from baseline at Day 14 | -0.06 (0.410) | -0.08 (0.422)
  Desquamation: At Baseline | 0.03 (0.164) | 0.05 (0.221)
  Desquamation: Change from baseline at 180 minutes | -0.03 (0.164) | -0.05 (0.221)
  Desquamation: Change from baseline at Day 1 | 0.08 (0.433) | 0.15 (0.533)
  Desquamation: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Desquamation: Change from baseline at Day 2 | 0.17 (0.507) | 0.18 (0.594)
  Desquamation: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Desquamation: Change from baseline at Day 3 | 0.17 (0.507) | 0.30 (0.648)
  Desquamation: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Desquamation: Change from baseline at Day 7 | 0.03 (0.291) | 0.05 (0.320)
  Desquamation: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Desquamation: Change from baseline at Day 14 | 0.00 (0.239) | -0.05 (0.223)
  Edema: At Baseline | 0.00 (0.00) | 0.03 (0.158)
  Edema: Change from baseline at 180 minutes | 0.00 (0.00) | -0.03 (0.158)
  Edema: Change from baseline at Day 1 | 0.03 (0.164) | -0.03 (0.158)
  Edema: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Edema: Change from baseline at Day 2 | 0.00 (0.00) | -0.03 (0.158)
  Edema: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Edema: Change from baseline at Day 3 | 0.00 (0.00) | -0.03 (0.158)
  Edema: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Edema: Change from baseline at Day 7 | 0.00 (0.00) | -0.03 (0.160)
  Edema: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Edema: Change from baseline at Day 14 | 0.00 (0.00) | -0.03 (0.160)

4. Secondary Outcome: Change From Baseline in Total Score of Participant Self-Assessment Scores
Description: Participant Self-Assessment was conducted by participants reflective of their skin condition at the time of evaluation. Participants scored following signs/symptom: pain, stinging/burning, itching, tightness, redness and dryness on scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Total score ranges as 0 to 18, higher score represents less tolerance to product applied.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
score on a scale
  At Baseline | 0.70 (1.024) | 1.15 (1.442)
  Change from baseline at 180 minutes | -0.43 (0.929) | -0.78 (1.250)
  Change from baseline at Day 1 | -0.24 (0.683) | -0.80 (1.506)
  Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 2 | -0.36 (0.762) | -0.43 (1.567)
  Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 3 | -0.50 (0.697) | -0.50 (1.485)
  Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 7 | -0.67 (0.894) | -0.85 (1.514)
  Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 14 | -0.61 (0.994) | -0.85 (1.631)

5. Secondary Outcome: Change From Baseline in Individual Participant Self-Assessment Scores for Pain, Stinging/Burning, Itching, Tightness, Redness and Dryness
Description: Participant Self-Assessment was conducted by participants reflective of their skin condition at the time of evaluation. Participants scored following signs/symptom: pain, stinging/burning, itching, tightness, redness and dryness on scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Higher score represents less tolerance to product applied.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
score on a scale
  Pain: At Baseline | 0.00 (0.00) | 0.00 (0.00)
  Pain: Change from baseline at 180 minutes | 0.00 (0.00) | 0.00 (0.00)
  Pain: Change from baseline at Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Pain: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Pain: Change from baseline at Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Pain: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Pain: Change from baseline at Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Pain: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Pain: Change from baseline at Day 7 | 0.00 (0.00) | 0.00 (0.00)
  Pain: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Pain: Change from baseline at Day 14 | 0.00 (0.00) | 0.00 (0.00)
  Stinging/Burning: At Baseline | 0.24 (0.548) | 0.43 (0.675)
  Stinging/Burning: Change from baseline at 180 min. | -0.19 (0.518) | -0.38 (0.628)
  Stinging/Burning: Change from baseline at Day 1 | -0.22 (0.534) | -0.43 (0.675)
  Stinging/Burning: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Stinging/Burning: Change from baseline at Day 2 | -0.25 (0.554) | -0.43 (0.675)
  Stinging/Burning: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Stinging/Burning: Change from baseline at Day 3 | -0.25 (0.554) | -0.43 (0.675)
  Stinging/Burning: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Stinging/Burning: Change from baseline at Day 7 | -0.25 (0.554) | -0.41 (0.677)
  Stinging/Burning: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Stinging/Burning: Change from baseline at Day 14 | -0.25 (0.554) | -0.41 (0.677)
  Itching: At Baseline | 0.00 (0.00) | 0.10 (0.379)
  Itching: Change from baseline at 180 min. | 0.00 (0.00) | -0.05 (0.316)
  Itching: Change from baseline at Day 1 | 0.03 (0.164) | -0.05 (0.450)
  Itching: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Itching: Change from baseline at Day 2 | 0.03 (0.167) | -0.03 (0.357)
  Itching: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Itching: Change from baseline at Day 3 | 0.06 (0.232) | -0.05 (0.450)
  Itching: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Itching: Change from baseline at Day 7 | 0.00 (0.00) | -0.08 (0.422)
  Itching: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Itching: Change from baseline at Day 14 | 0.00 (0.00) | -0.10 (0.384)
  Tightness: At Baseline | 0.00 (0.00) | 0.08 (0.267)
  Tightness: Change from baseline at 180 min. | 0.00 (0.00) | -0.05 (0.221)
  Tightness: Change from baseline at Day 1 | 0.05 (0.329) | -0.03 (0.357)
  Tightness: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Tightness: Change from baseline at Day 2 | 0.06 (0.232) | 0.05 (0.389)
  Tightness: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Tightness: Change from baseline at Day 3 | 0.00 (0.00) | 0.05 (0.389)
  Tightness: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Tightness: Change from baseline at Day 7 | 0.00 (0.00) | -0.05 (0.223)
  Tightness: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Tightness: Change from baseline at Day 14 | 0.00 (0.00) | -0.03 (0.280)
  Redness: At Baseline | 0.32 (0.530) | 0.40 (0.672)
  Redness: Change from baseline at 180 min. | -0.11 (0.516) | -0.20 (0.648)
  Redness: Change from baseline at Day 1 | -0.16 (0.501) | -0.38 (0.667)
  Redness: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Redness: Change from baseline at Day 2 | -0.33 (0.535) | -0.33 (0.730)
  Redness: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Redness: Change from baseline at Day 3 | -0.33 (0.535) | -0.33 (0.730)
  Redness: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Redness: Change from baseline at Day 7 | -0.33 (0.535) | -0.38 (0.673)
  Redness: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Redness: Change from baseline at Day 14 | -0.33 (0.535) | -0.33 (0.737)
  Dryness: At Baseline | 0.14 (0.347) | 0.15 (0.362)
  Dryness: Change from baseline at 180 min. | -0.14 (0.347) | -0.10 (0.304)
  Dryness: Change from baseline at Day 1 | 0.05 (0.405) | 0.08 (0.526)
  Dryness: Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Dryness: Change from baseline at Day 2 | 0.14 (0.424) | 0.30 (0.648)
  Dryness: Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Dryness: Change from baseline at Day 3 | 0.03 (0.446) | 0.25 (0.543)
  Dryness: Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Dryness: Change from baseline at Day 7 | -0.08 (0.280) | 0.08 (0.580)
  Dryness: Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Dryness: Change from baseline at Day 14 | -0.03 (0.506) | 0.03 (0.486)

6. Secondary Outcome: Change From Baseline in Trans-epidermal Water Loss (TEWL)
Description: Trans-epidermal water loss (TEWL) measurement was performed by evaporimetry with a Tewameter to assess skin barrier function. Measurements was done in triplicate on the left cheek (below the cheekbone between the nose and ear). TEWL measurements was performed the participant lying horizontally, on their back, so that the chimney of the Tewameter probe was aligned vertically.
Time Frame: At baseline (60 mins. post procedure but prior to any test product application) and 180 mins, 360 mins, 1 day, 2 days, 3 days, 7 days and 14 days after completion of the facial peel procedure
Population: Intent-to-treat (ITT) population included all randomized participants. Number of participants analyzed are the part of ITT population analyzed for this outcome at specific time points.
Measure: Mean (Standard Deviation); unit: gram per square meter per hour (g/m2/hr)
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
gram per square meter per hour (g/m2/hr)
  At Baseline | 20.20 (5.158) | 20.24 (5.242)
  Change from baseline at 180 min. | 0.50 (1.940) | 0.32 (1.818)
  Change from baseline at 360 min.: number analyzed (Participants) | 37 | 39
  Change from baseline at 360 min. | -0.47 (2.803) | -0.72 (2.729)
  Change from baseline at Day 1: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 1 | -0.83 (2.958) | -0.76 (2.567)
  Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 2 | -1.38 (2.782) | -1.22 (3.182)
  Change from baseline at Day 3: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 3 | -1.27 (2.886) | -0.05 (3.644)
  Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 7 | -2.39 (3.263) | -0.65 (4.552)
  Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 14 | -2.92 (3.028) | -1.64 (4.329)

7. Secondary Outcome: Change From Baseline in Corneometer Measurements
Description: Corneometry was used to measure moisture content of stratum corneum using corneometer. The corneometer probe was placed in contact with the skin of the participant's test site for 1-2 s per measurement. The corneometer measurements were performed in triplicate at the left cheek (below the cheekbone, between the nose and ear) with the participant lying horizontally, on their back. Corneometer values were measured at 180 mins, 360 mins, 1 day, 2 days, 3 days, 7 days and 14 days after completion of the facial peel procedure to evaluate the impact of twice-daily application of the investigational products on skin moisturization compared to the use of no test product. An increase in Corneometer values corresponds to skin-moisturizing effect.
Time Frame: as for outcome 6
Population: ITT population included all randomized participants. Number of participants analyzed are the part of ITT population analyzed for this outcome at specific time points.
Measure: Mean (Standard Deviation); unit: corneometer units
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
corneometer units
  At Baseline | 67.17 (11.017) | 69.17 (11.635)
  Change from baseline at 180 min. | 13.93 (9.919) | -2.30 (6.388)
  Change from baseline at 360 min. | 9.55 (9.915) | -1.96 (7.581)
  Change from baseline at Day 1 | -2.00 (8.178) | -9.75 (9.051)
  Change from baseline at Day 2: number analyzed (Participants) | 36 | 40
  Change from baseline at Day 2 | -2.03 (9.776) | -9.42 (9.349)
  Change from baseline at Day 3: number analyzed (Participants) | 35 | 40
  Change from baseline at Day 3 | -0.36 (7.909) | -6.61 (10.125)
  Change from baseline at Day 7: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 7 | -3.22 (8.232) | -10.28 (10.967)
  Change from baseline at Day 14: number analyzed (Participants) | 36 | 39
  Change from baseline at Day 14 | -0.91 (8.413) | -9.18 (10.167)

8. Other Pre Specified Outcome: Number of Participants With Global Self-Assessment of Satisfaction Score
Description: Participants rated the level of satisfaction with the post-procedure skin care regimen to which they were randomized using scale as follows: 0 (Very satisfied), 1 (Satisfied), 2 (Poorly satisfied), 3 (Not at all satisfied).
Time Frame: 14 days after completion of the facial peel procedure
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
Number analyzed (Participants) | 37 | 40
Participants
  Missing | 1 | 1
  Very Satisfied | 17 | 12
  Satisfied | 19 | 26
  Poorly Satisfied | 0 | 1
  Not at all Satisfied | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 26 days (from Visit 1 to until 5 days following last administration on Visit 8)
Arm/Group | Group 1 (Test Product) | Group 2 (No Test Product)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/40
Other Adverse Events (participants affected / at risk) | 1/37 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Test Product) (N=37) | Group 2 (No Test Product) (N=40)
Scab (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03103906/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT03103906/SAP_001.pdf